CLINICAL TRIAL: NCT03683160
Title: A Cognitive-Augmented Mobility Program (CAMP): Combining Cognitive Strategy Training And Best Evidence Mobility Training To Optimize Long-Term Meaningful Living For People With Stroke
Brief Title: A Cognitive-Augmented Mobility Program
Acronym: CAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 446-2016
Record Dates: First submitted 2018-09-05; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: Stroke, mobility, cognitive strategy training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single arm design with two blocks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Augmented Mobility Program (Experimental): CAMP will combine education, one-on-one cognitive strategy training, and a cardiovascular and strength-training program conducted within a group setting. It will be run as a group of up to 6 participants, facilitated by a physiotherapist and a physiotherapy assistant or kinesiologist. It consists of 2 phases with a total of 19 sessions: Intervention Preparation (3 sessions), Active Intervention (16 sessions), and Follow-Up (1 session).
  Interventions: Other: Cognitive Augmented Mobility Program

INTERVENTIONS:
Other: Cognitive Augmented Mobility Program — CAMP will combine education, one-on-one cognitive strategy training, and a cardiovascular and strength-training program conducted within a group setting. It will be run as a group of up to 6 participants, facilitated by a physiotherapist and a physiotherapy assistant or kinesiologist. It consists of 2 phases with a total of 19 sessions: Intervention Preparation (3 sessions), Active Intervention (16 sessions), and Follow-Up (1 session).

SUMMARY:
This project will combine best-evidence gait and mobility training with best evidence cognitive strategy training to produce a new cognitive-augmented mobility intervention that is expected to optimize long-term functional mobility outcomes for those living with stroke. More importantly, the new cognitive-augmented mobility program (CAMP) will address two crucial outcomes that do not occur with current approaches: 1. Maintenance of mobility gains after discharge from formal rehabilitation and 2. Transfer of skills learned in rehabilitation to real-world community living. This project will result in a new, fully defined intervention, and will provide effect size and cost estimates to design a future appropriately powered randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Difficulty walking is a leading cause of activity restriction in survivors of stroke. It is directly related to important functional issues, such as challenges in crossing a street in time, difficulty walking to a bus stop and increased risk of falls. These functional issues can then impact a person's confidence to move around their community, ultimately leading to lower levels of physical activity and potential negative health consequences. The best way to optimize recovery in walking and mobility is not yet known, and there are critical gaps in existing treatments. While some approaches are effective in the short term, strategies to promote the maintenance of improvements are not well established, benefits are usually not transferred beyond the specific skills trained and the specific context in which they were learned, few interventions impact community participation, and cost effectiveness has rarely been investigated. A potential solution exists in combining best-evidence interventions: task-specific gait and mobility training to improve skill quality, cardiorespiratory and strength exercises to improve endurance and speed, and cognitive strategy training to teach problem solving, improve confidence and to ensure long-term maintenance and transfer of skills to home and community settings. The investigators will combine best evidence mobility interventions with best evidence cognitive strategy training to develop and evaluate a new intervention to optimize long-term functional mobility outcomes for those living with stroke. The project consists of two sequential stages: 1) intervention development through literature synthesis; face validity testing using focus groups with patients, family members and expert stroke rehabilitation clinicians; and intervention refinement; followed by 2) feasibility/pilot testing with 10 people more than 6 months post stroke. Anticipated outcomes include a fully developed intervention with the potential to optimize mobility rehabilitation and effect size estimates to permit the design of a future, appropriately-powered randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years of age or older
* post stroke
* have completed outpatient therapy
* can walk a minimum of 3 metres with or without an aid

Exclusion Criteria:

* patient does not a mobility goal
* neurological diagnoses other than stroke
* major psychiatric illness
* significant dementia (MoCA scores < 21)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Mean Canadian Occupational Performance Measure scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  The Canadian Occupational Performance Measure (COPM) is a self-report measure of performance and satisfaction with self-selected goals. Participants are asked to generate 5 personally meaningful rehabilitation goals and rate their current performance and satisfaction on a scale from 1 to 10. Total scores are the average performance and satisfaction score. Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
Mean 5 metre walk test scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  Measure of gait speed in metres per second. Higher scores indicate faster walking speed.
Mean 6-minute walk test scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  Measure of walking endurance in metres walked. Higher scores indicate greater distance traveled.
Mean Berg Balance Scale scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  The Berg Balance Scale (BBS) is a measure of static balance. Participants are asked to complete a series of 14 tasks and are scored from 0 to 4. Total score (min=0; max=56) is calculated by adding the scores of the individual tasks, higher scores indicate better outcomes.
Mean Activity-specific Balance Confidence Scale scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  The Activity-specific Balance Confidence (ABC) Scale is a self-report measure of confidence to perform daily activities without falling. Participants assign a score from 0 to 100 to each of the measure's 16 items and the total score is calculated by obtaining the average score. Higher scores indicate better outcomes.
Mean Community Balance and Mobility Scale scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  The Community Balance and Mobility (CB&M) Scale is a measure of balance and mobility. Participants are asked to perform 13 tasks while a therapist scores their performance. Several tasks require using both sides. The total score (min=0; max=96) is the sum of all task scores and greater scores indicate better outcomes.
Mean Functional Independence Measure scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  The Functional Independence Measure (FIM) is a measure of the amount of assistance required to complete activities of daily living. Participants are asked about the amount of assistance required to complete each of the measure's 18 items and are assigned a score from 1 to 7 for each item. Total scores (min=18; max=126) are the sum of the item scores and greater scores indicate better outcomes.
Mean Stroke Impact Scale scores | 1) 1 week pre-intervention; 2) 1 week post-intervention, 3) 4 to 5 weeks post-intervention
  The Stroke Impact Scale (SIS) is a self-report measure of perceived impact of stroke on function and everyday life. The SIS is a 56 item measure with 8 subscales measuring strength, hand function, ADL/IADL, mobility, communication, emotion, memory and thinking, and participation/role function. Subscale scores range from 0 to 100. Greater scores indicate better outcomes.

OTHER OUTCOMES:
Acceptability - Participant satisfaction and intent to use | 1 week post-intervention
  Participants will be asked to complete a 2 question survey to gauge their satisfaction with the intervention and their interest in using the skills they learned during the intervention. Scores for each item range from 1 to 5. Higher scores indicate greater satisfaction and intention to use the skills they learned in the future.
Feasibility - Number of participants recruited | Through study completion, up to 9 months
  Total number of participants enrolled in the study
Feasibility - Number of participants who attend the intervention session | Through study completion, up to 9 months
  Total number of participants who attend the intervention sessions
Feasibility - Number of participant withdrawals | Through study completion, up to 9 months
  Number of participant withdrawals and reasons, if any
Feasibility - Number of adverse events | Through study completion, up to 9 months
  Total number of adverse events and reasons, if any

CONTACTS AND LOCATIONS:
Overall Officials: Sara McEwen, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, St. John's Rehab, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/60/NCT03683160/Prot_000.pdf